CLINICAL TRIAL: NCT00985621
Title: A PHASE 3 RANDOMIZED, DOUBLE-BLIND, PLACEBO AND OXYCODONE CONTROLLED MULTI-CENTER STUDY OF THE EFFICACY AND SAFETY OF TANEZUMAB IN PATIENTS WITH OSTEOARTHRITIS OF THE KNEE OR HIP
Brief Title: Tanezumab In Osteoarthritis Of The Hip Or Knee
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A4091030; 2009-013329-41 (EudraCT Number); OA OXY STUDY (Other: Alias Study Number)
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Results first posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis
Keywords: monoclonal antibody; RN624; PF-04383119; nerve growth factor; OA; pain; arthritis
MeSH Terms: conditions — Osteoarthritis; Hereditary Sensory and Autonomic Neuropathies; Pain; Arthritis | interventions — tanezumab; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental)
  Interventions: Biological: tanezumab 10 mg
- 2 (Experimental)
  Interventions: Biological: tanezumab 5 mg
- 3 (Active Comparator)
  Interventions: Drug: oxycodone
- 4 (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Biological: tanezumab 10 mg — tanezumab 10 mg one dose at weeks 0 and 8
  Arms: 1
Biological: tanezumab 5 mg — tanezumab 5 mg one dose at weeks 0 and 8
  Arms: 2
Drug: oxycodone — oxycodone CR, 10-40 mg q12h
  Arms: 3
Other: placebo — placebo
  Arms: 4

SUMMARY:
The purpose of the study is to test the efficacy and safety of 2 doses of tanezumab compared to oxycodone CR and placebo in patients with osteoarthritis

DETAILED DESCRIPTION:
This study was terminated on 13 Dec 2010 following a US FDA clinical hold for tanezumab osteoarthritis clinical studies which halted dosing and enrollment of patients on 23 June 2010 for potential safety issues.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis of the knee or hip according to Kellgren-Lawrence x-ray grade of 2

Exclusion Criteria:

* pregnancy or intent to become pregnant
* BMI greater than 39
* other severe pain, significant cardiac, neurological or psychiatric disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2009-10-30 (Actual); Primary Completion 2010-12-13 (Actual); Study Completion 2011-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (108):
- United States (64):
  - Achieve Clinical Research, Birmingham, Alabama
  - Alabama Orthopaedic Clinics, PC, Mobile, Alabama
  - Horizon Research Group, Inc., Mobile, Alabama
  - Arizona Research Center, Inc., Phoenix, Arizona
  - Osteoporosis Medical Center, Beverly Hills, California
  - Med Frontier Clinical Research, Buena Park, California
  - Providence Clinical Research, Burbank, California
  - Valley Research, Fresno, California
  - Apex Research Institute, Santa Ana, California
  - Medvin Clinical Research, Van Nuys, California
  - Advanced Radiology, Stamford, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Clinical Research of South Florida, Coral Gables, Florida
  - Homestead Clinical Research Group, P.A., Cutler Bay, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Florida Clinical Research Center, LLC, Fruitland Park, Florida
  - Adult Medicine Specialists, Longwood, Florida
  - Genesis Research International, Longwood, Florida
  - Community Research Foundation, Inc., Miami, Florida
  - Compass Research, LLC, Orlando, Florida
  - Advent Clinical Research Centers, Inc., Pinellas Park, Florida
  - Sarasota Center For Clinical Research, Sarasota, Florida
  - Dale G. Bramlet, MD, St. Petersburg, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Laureate Clinical Research Group, Atlanta, Georgia
  - Drug Studies America Inc., Marietta, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - North Goergia Internal Medicine, Woodstock, Georgia
  - Americana Orthopedics, Boise, Idaho
  - Sonora Clinical Research, LLC., Boise, Idaho
  - Northwest Indiana Center for Clinical Research, Valparaiso, Indiana
  - Commonwealth Biomedical Research, Madisonville, Kentucky
  - Mid-Atlantic Medical Research, Hollywood, Maryland
  - Miray Medical Center, Brockton, Massachusetts
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Great Lakes Research Group, Incorporated, Bay City, Michigan
  - The Center for Clinical Trials, Biloxi, Mississippi
  - Mercy Health Research, St Louis, Missouri
  - Midwest Minor Medical, Omaha, Nebraska
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Diagnostic Center of Medicine, Henderson, Nevada
  - Office of Matthew Barton, MD, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Office of Andrew J. Porges, MD PC, Roslyn, New York
  - MediSpect, LLC, Boone, North Carolina
  - Crescent Medical Research, Salisbury, North Carolina
  - Hilltop Medical Research Center, Cincinnati, Ohio
  - Columbus Clinical Research, Columbus, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Piedmont Arthritis Clinic, PA, Greenville, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - TriCities Medical Research, Bristol, Tennessee
  - Appalachian Medical Research Inc., Johnson City, Tennessee
  - ClinRx Research, LLC, Carrollton, Texas
  - Tekton Research, Inc, Georgetown, Texas
  - One Step Diagnostic (X-Ray Facility), Houston, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Leander Healthcare Center, Leander, Texas
  - ClinRx Research, Richardson, Texas
  - Oakwell Clinical research, LLC, San Antonio, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
- Austria (5):
  - LKH/Universitatsklinikum Graz, Graz
  - Nuhr Zentrum, Senftenberg
  - ClinPharm International GmbH, Vienna
  - Synexus ClinPharm GmbH, Vienna
  - Rheuma Zentrum Favoriten, Vienna
- Denmark (4):
  - CCBR A/S, Aalborg
  - CCBR A/S, Ballerup Municipality
  - Frederiksberg Hospital Parker Institute, Frederiksberg
  - CCBR A/S, Vejle
- Germany (21):
  - Charité Universitätsmedizin Berlin, Berlin
  - Klinische Forschung Berlin-Buch GmbH, Berlin
  - Viereck-Apotheke, Berlin
  - Charité Campus Virchow-Klinikum Apotheke, Berlin
  - ClinPharm International GmbH, Bochum
  - Herz Apotheke, Bochum
  - Synexus ClinPharm GmbH, Bochum
  - Synexus ClinPharm GmbH / Frankfurt/M, Frankfurt am Main
  - Schiller-Apotheke, Göppingen
  - Schmerz und Palliativ-Zentrum Goppingen, Göppingen
  - Falken Apotheke Hoheluft, Hamburg
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Klinische Forschung Hannover-Mitte GmbH, Hanover
  - Löwen Apotheke, Hanover
  - Synexus ClinPharm GmbH, Leipzig
  - Arkana Apotheke OHG, Leipzig
  - Synexus ClinPharm GmbH Pruefzentrum Magdeburg, Magdeburg
  - Apotheke im MSZ, Magdeburg
  - Schwanen Apotheke am Markt, Offenbach
  - Klinische Forschung Schwerin GmbH, Schwerin
  - Sonnenapotheke, Schwerin
- Poland (6):
  - Nzoz Centrum Medyczne, Bialystok
  - Szpital Specjalistyczny im. J. Dietla, Krakow
  - NZOZ REUMED Sp.zo.o., Lublin
  - Medyczne Centrum Hetmanska, Poznan
  - NZOZ "Nasz Lekarz", Torun
  - Centrum Medyczne OSTEOMED NZOZ, Warsaw
- Spain (4):
  - Hospital Nuestra Senora de la Esperanza, Santiago de Compostela, A Coruña
  - Complejo Hospitalario Universitario de A Coruna, A Coruña
  - Hospital Regional Universitario Carlos Haya (Hospital Civil), Málaga
  - Hospital Universitario Virgen Macarena, Seville
- Sweden (4):
  - Me3plus AB, Gothenburg
  - Avdelningen for klinisk provning, Sahlgrenska Universitetssjukhuset, Gothenburg
  - Center for Clinical Studies, Malmo
  - Bragee Medect AB, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Brown MT, Cornblath DR, Koltzenburg M, Gorson KC, Hickman A, Pixton GC, Gaitonde P, Viktrup L, West CR. Peripheral Nerve Safety of Nerve Growth Factor Inhibition by Tanezumab: Pooled Analyses of Phase III Clinical Studies in Over 5000 Patients with Osteoarthritis. Clin Drug Investig. 2023 Jul;43(7):551-563. doi: 10.1007/s40261-023-01286-3. Epub 2023 Jul 18. PMID 37460782
- [Derived] Tive L, Bello AE, Radin D, Schnitzer TJ, Nguyen H, Brown MT, West CR. Pooled analysis of tanezumab efficacy and safety with subgroup analyses of phase III clinical trials in patients with osteoarthritis pain of the knee or hip. J Pain Res. 2019 Mar 19;12:975-995. doi: 10.2147/JPR.S191297. eCollection 2019. PMID 30936738
- [Derived] Spierings ELH, Fidelholtz J, Wolfram G, Smith MD, Brown MT, West CR. A phase III placebo- and oxycodone-controlled study of tanezumab in adults with osteoarthritis pain of the hip or knee. Pain. 2013 Sep;154(9):1603-1612. doi: 10.1016/j.pain.2013.04.035. Epub 2013 Apr 22. PMID 23707270
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091030&StudyName=Tanezumab%20In%20Osteoarthritis%20Of%20The%20Hip%20Or%20Knee

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to tanezumab (RN624 or PF-04383119) intravenous (IV) infusion over 5 minutes on Day 1 and Week 8, along with placebo matched to oxycodone controlled released (CR) tablet orally twice daily up to Week 16.
- Tanezumab 5 mg: Tanezumab (RN624 or PF-04383119) 5 milligram (mg) intravenous infusion over 5 minutes on Day 1 and Week 8, along with placebo matched to oxycodone CR tablet orally twice daily up to Week 16.
- Tanezumab 10 mg: Tanezumab (RN624 or PF-04383119) 10 mg intravenous infusion over 5 minutes on Day 1 and Week 8, along with placebo matched to oxycodone CR tablet orally twice daily up to Week 16.
- Oxycodone CR: Placebo matched to tanezumab (RN624 or PF-04383119) intravenous infusion over 5 minutes on Day 1 and Week 8, along with oxycodone CR tablet at a starting dose of 10 mg orally twice daily up to Week 16. Oxycodone dose was adjusted according to the pain relief and tolerability up to a maximum of 40 mg orally twice daily.
Period: Overall Study
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Started | 142 | 161 | 152 | 159
Treated | 141 | 161 | 150 | 158
Completed | 28 | 30 | 29 | 22
Not Completed | 114 | 131 | 123 | 137
Not completed — Adverse Event | 2 | 3 | 4 | 16
Not completed — Lack of Efficacy | 10 | 6 | 5 | 12
Not completed — Lost to Follow-up | 2 | 3 | 4 | 4
Not completed — Study Terminated by Sponsor | 89 | 108 | 99 | 92
Not completed — Protocol Violation | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 8 | 10 | 8 | 12
Not completed — Other | 1 | 0 | 0 | 0
Not completed — Randomized but not Treated | 1 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all randomized participants who received at least 1 dose of randomized intravenous study medication (either tanezumab or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR | Total
Number analyzed (Participants) | 141 | 161 | 150 | 158 | 610
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (10.5) | 57.8 (9.2) | 57.0 (9.8) | 57.6 (9.1) | 57.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 96 | 94 | 99 | 381
  Male | 49 | 65 | 56 | 59 | 229

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 8: ITT Population
Description: The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis (OA) in the index joint (knee/hip) during past 48 hours. It is calculated as the mean of the scores from the 5 individual questions scored on a numerical rating scale (NRS) of 0 to 10, where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 to 10, where higher scores indicate higher pain.
Time Frame: Baseline, Week 8
Population: ITT analysis set included all randomized participants who received at least 1 dose of randomized intravenous study medication (either tanezumab or placebo). Missing data were imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
units on a scale
  Baseline | 7.75 (1.21) | 7.85 (1.27) | 7.63 (1.30) | 7.85 (1.27)
  Change at Week 8 | -2.74 (2.26) | -3.71 (2.49) | -3.63 (2.62) | -2.71 (2.36)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg; Analysis was performed using analysis of co-variance (ANCOVA) model with treatment as main effect, baseline value, index joint, previous opioid use as covariates, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA; Least Squares (LS) Mean Difference = -0.96, 95% CI 2-sided [-1.49 to -0.44], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.97, 95% CI 2-sided [-1.50 to -0.43], Standard Error of Mean 0.27

2. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 8: Modified Intent-to-Treat (mITT) Population
Description: The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to OA in the index joint (knee/hip) during past 48 hours. It is calculated as the mean of the scores from the 5 individual questions scored on an NRS of 0 to 10, where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 to 10, where higher scores indicate higher pain.
Time Frame: Baseline, Week 8
Population: Modified intent-to-treat (mITT) analysis set included all participants in ITT analysis set who had Week 8 visit on or before 23 June 2010 (effective date of the United States Food and Drug Administration [US FDA] imposed clinical hold). Missing data were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 137 | 153 | 149 | 156
units on a scale
  Baseline | 7.75 (1.20) | 7.87 (1.26) | 7.64 (1.31) | 7.86 (1.27)
  Change at Week 8 | -2.58 (2.30) | -3.42 (2.64) | -3.01 (2.69) | -2.41 (2.29)
Statistical Analysis 1: Comparison: Tanezumab 5 mg vs Oxycodone CR; Analysis was performed using ANCOVA model with treatment as main effect, baseline value, index joint, previous opioid use as covariates, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.97, 95% CI 2-sided [-1.49 to -0.45], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: Tanezumab 10 mg vs Oxycodone CR; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.018, ANCOVA; LS Mean Difference = -0.63, 95% CI 2-sided [-1.16 to -0.11], Standard Error of Mean 0.27
Statistical Analysis 3: Comparison: Placebo vs Oxycodone CR; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.700, ANCOVA; LS Mean Difference = 0.11, 95% CI 2-sided [-0.43 to 0.65], Standard Error of Mean 0.28

3. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Weeks 2, 4, 12, and 16: ITT Population
Description: as for outcome 2
Time Frame: Baseline, Weeks 2, 4, 12, and 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of randomized intravenous study medication (either tanezumab or placebo). Missing data were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
units on a scale
  Change at Week 2 | -2.12 (1.91) | -2.47 (2.23) | -2.29 (2.25) | -2.31 (2.09)
  Change at Week 4 | -2.55 (2.09) | -3.56 (2.54) | -3.45 (2.62) | -2.87 (2.25)
  Change at Week 12 | -2.85 (2.37) | -3.82 (2.62) | -3.64 (2.60) | -2.80 (2.41)
  Change at Week 16 | -2.95 (2.46) | -3.80 (2.60) | -3.65 (2.51) | -2.79 (2.39)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg; Change at Week 2: analysis was performed using ANCOVA model with treatment as main effect, baseline value, index joint, previous opioid use as covariates, and study site as a random effect; Test type: Superiority or Other; p = 0.177, ANCOVA; LS Mean Difference = -0.32, 95% CI 2-sided [-0.78 to 0.14], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.416, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-0.66 to 0.28], Standard Error of Mean 0.24
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 5 mg; Change at Week 4: analysis was performed using ANCOVA model with treatment as main effect, baseline value, index joint, previous opioid use as covariates, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.98, 95% CI 2-sided [-1.50 to -0.46], Standard Error of Mean 0.26
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.95, 95% CI 2-sided [-1.48 to -0.43], Standard Error of Mean 0.27

4. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Weeks 2, 4, 12, and 16: mITT Population
Description: as for outcome 2
Time Frame: Baseline, Weeks 2, 4, 12, and 16
Population: mITT analysis set included all participants in ITT analysis set who had Week 8 visit on or before 23 June 2010 (effective date of the US FDA imposed clinical hold). Missing data were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 137 | 153 | 149 | 156
units on a scale
  Change at Week 2 | -1.98 (1.92) | -2.34 (2.25) | -2.05 (2.18) | -2.08 (2.17)
  Change at Week 4 | -2.37 (2.15) | -3.27 (2.58) | -2.85 (2.68) | -2.48 (2.29)
  Change at Week 12 | -2.69 (2.42) | -3.58 (2.76) | -3.06 (2.69) | -2.57 (2.37)
  Change at Week 16 | -2.85 (2.55) | -3.63 (2.77) | -3.16 (2.68) | -2.58 (2.35)
Statistical Analysis 1: Comparison: Tanezumab 5 mg vs Oxycodone CR; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.319, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.69 to 0.22], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Tanezumab 10 mg vs Oxycodone CR; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.916, ANCOVA; LS Mean Difference = 0.02, 95% CI 2-sided [-0.43 to 0.48], Standard Error of Mean 0.23
Statistical Analysis 3: Comparison: Placebo vs Oxycodone CR; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.526, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.63 to 0.32], Standard Error of Mean 0.24
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs Oxycodone CR; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.004, ANCOVA; LS Mean Difference = -0.75, 95% CI 2-sided [-1.26 to -0.24], Standard Error of Mean 0.26
Statistical Analysis 5: Comparison: Tanezumab 10 mg vs Oxycodone CR; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.134, ANCOVA; LS Mean Difference = -0.39, 95% CI 2-sided [-0.90 to 0.12], Standard Error of Mean 0.26
Statistical Analysis 6: Comparison: Placebo vs Oxycodone CR; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.497, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.71 to 0.35], Standard Error of Mean 0.27

5. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale Score at Weeks 2, 4, 8, 12, and 16: ITT Population
Description: The WOMAC physical function subscale is a 17-item questionnaire used to assess the degree of difficulty experienced due to OA in the index joint (knee/hip) during past 48 hours. It is calculated as the mean of the scores from the 17 individual questions scored on an NRS of 0 to 10, where higher scores indicate worse function. Total score range for WOMAC physical function subscale score is 0 to 10, where higher scores indicate worse function. Physical function refers to participant's ability to move around and perform usual activities of daily living.
Time Frame: Baseline, Week 2, 4, 8, 12, and 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of randomized intravenous study medication (either tanezumab or placebo). Missing data were imputed using LOCF. Here 'overall number of participants analyzed' signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 140 | 161 | 150 | 158
units on a scale
  Baseline | 7.19 (1.50) | 7.30 (1.58) | 7.04 (1.54) | 7.25 (1.53)
  Change at Week 2 | -1.51 (1.73) | -2.16 (2.30) | -1.95 (2.08) | -1.71 (1.94)
  Change at Week 4 | -1.89 (1.96) | -3.04 (2.59) | -2.94 (2.61) | -2.10 (2.20)
  Change at Week 8 | -2.01 (2.09) | -3.18 (2.49) | -3.08 (2.50) | -2.14 (2.30)
  Change at Week 12 | -2.17 (2.26) | -3.34 (2.62) | -3.09 (2.45) | -2.17 (2.28)
  Change at Week 16 | -2.26 (2.37) | -3.27 (2.61) | -3.10 (2.42) | -2.18 (2.26)

6. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale Score at Weeks 2, 4, 8, 12, and 16: mITT Population
Description: as for outcome 5
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: mITT analysis set included all participants in ITT analysis set who had Week 8 visit on or before 23 June 2010 (effective date of the US FDA imposed clinical hold). Missing data were imputed using LOCF. Here 'overall number of participants analyzed' signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 136 | 153 | 149 | 156
units on a scale
  Baseline | 7.17 (1.51) | 7.32 (1.59) | 7.05 (1.54) | 7.26 (1.53)
  Change at Week 2 | -1.41 (1.73) | -2.00 (2.32) | -1.73 (1.99) | -1.56 (1.94)
  Change at Week 4 | -1.73 (2.00) | -2.80 (2.69) | -2.47 (2.59) | -1.83 (2.16)
  Change at Week 8 | -1.87 (2.03) | -3.00 (2.68) | -2.62 (2.58) | -1.87 (2.24)
  Change at Week 12 | -2.03 (2.21) | -3.19 (2.78) | -2.65 (2.60) | -1.95 (2.24)
  Change at Week 16 | -2.20 (2.38) | -3.22 (2.78) | -2.77 (2.64) | -1.97 (2.21)

7. Secondary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Osteoarthritis at Weeks 2, 4, 8, 12, and 16: ITT Population
Description: PGA: Participants answered the following question: "Considering all the ways the OA in your index (knee/hip) affects you, how are you doing today?" Participants rated their condition by using a 5-point Likert scale: 1) very good (asymptomatic and no limitation of normal activities); 2) good (mild symptoms and no limitation of normal activities); 3) fair (moderate symptoms and limitation of some normal activities); 4) poor (severe symptoms and inability to carry out most normal activities); and 5) very poor (very severe symptoms which are intolerable and inability to carry out all normal activities). Higher score indicated severe condition.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
units on a scale
  Baseline | 3.60 (0.68) | 3.58 (0.65) | 3.57 (0.68) | 3.59 (0.62)
  Change at Week 2 | -0.49 (0.88) | -0.71 (0.90) | -0.63 (0.78) | -0.54 (0.76)
  Change at Week 4 | -0.57 (0.85) | -0.99 (0.96) | -0.99 (0.84) | -0.64 (0.78)
  Change at Week 8 | -0.56 (0.86) | -0.93 (0.97) | -1.01 (0.97) | -0.58 (0.78)
  Change at Week 12 | -0.64 (0.88) | -0.99 (0.97) | -1.07 (0.96) | -0.59 (0.86)
  Change at Week 16 | -0.63 (0.87) | -0.96 (0.97) | -1.07 (0.95) | -0.59 (0.83)

8. Secondary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Osteoarthritis at Weeks 2, 4, 8, 12, and 16: mITT Population
Description: as for outcome 7
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 137 | 153 | 149 | 156
units on a scale
  Baseline | 3.59 (0.68) | 3.59 (0.65) | 3.56 (0.68) | 3.59 (0.62)
  Change at Week 2 | -0.47 (0.88) | -0.71 (0.89) | -0.55 (0.76) | -0.49 (0.74)
  Change at Week 4 | -0.50 (0.86) | -0.94 (0.95) | -0.82 (0.82) | -0.54 (0.75)
  Change at Week 8 | -0.55 (0.91) | -0.93 (0.98) | -0.81 (0.84) | -0.52 (0.74)
  Change at Week 12 | -0.63 (0.93) | -0.98 (0.96) | -0.83 (0.84) | -0.56 (0.81)
  Change at Week 16 | -0.67 (0.94) | -0.97 (0.97) | -0.87 (0.83) | -0.55 (0.79)

9. Secondary Outcome: Number of Participants With Outcome Measures in Rheumatology - Osteoarthritis Research Society International (OMERACT-OARSI) Response at Weeks 2, 4, 8, 12, and 16: ITT Population
Description: OMERACT-OARSI response: greater than or equal to (>=) 50 percent (%) improvement from baseline and absolute change from baseline of >=2 units at Week of interest in WOMAC pain or physical function subscales, or at least 2 of the following 3 being true: >=20% improvement from baseline and absolute change from baseline of >=1 unit at Week of interest in 1) WOMAC pain subscale, 2) WOMAC physical function subscale, 3) PGA of osteoarthritis (score: 1-5, higher score=more affected). WOMAC pain, physical function subscales assess amount of pain/difficulty experienced (score: 0-10, higher score=higher pain/difficulty).
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
Participants
  Week 2 | 70 | 89 | 82 | 81
  Week 4 | 87 | 117 | 107 | 97
  Week 8 | 81 | 120 | 105 | 93
  Week 12 | 83 | 120 | 110 | 100
  Week 16 | 84 | 120 | 112 | 95

10. Secondary Outcome: Number of Participants With Outcome Measures in Rheumatology - Osteoarthritis Research Society International (OMERACT-OARSI) Response at Weeks 2, 4, 8, 12, and 16: mITT Population
Description: OMERACT-OARSI response: >=50 percent (%) improvement from baseline and absolute change from baseline of >=2 units at Week of interest in WOMAC pain or physical function subscales, or at least 2 of the following 3 being true: >=20% improvement from baseline and absolute change from baseline of >=1 unit at Week of interest in 1) WOMAC pain subscale, 2) WOMAC physical function subscale, 3) PGA of osteoarthritis (score: 1-5, higher score=more affected). WOMAC pain, physical function subscales assess amount of pain/difficulty experienced (score: 0-10, higher score=higher pain/difficulty).
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 137 | 153 | 149 | 156
Participants
  Week 2 | 64 | 79 | 74 | 70
  Week 4 | 76 | 105 | 87 | 83
  Week 8 | 78 | 108 | 86 | 80
  Week 12 | 80 | 110 | 89 | 87
  Week 16 | 84 | 111 | 93 | 87

11. Secondary Outcome: Number of Participants With At Least (>=) 30 Percent (%), 50%, 70% and 90% Reduction From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Weeks 2, 4, 8, 12, and 16: ITT Population
Description: as for outcome 2
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
Participants
  Week 2: >=30% Reduction | 59 | 75 | 66 | 71
  Week 2: >=50% Reduction | 30 | 46 | 42 | 33
  Week 2: >=70% Reduction | 10 | 23 | 15 | 13
  Week 2: >=90% Reduction | 1 | 5 | 4 | 5
  Week 4: >=30% Reduction | 72 | 98 | 97 | 86
  Week 4: >=50% Reduction | 44 | 72 | 68 | 48
  Week 4: >=70% Reduction | 15 | 48 | 47 | 25
  Week 4: >=90% Reduction | 3 | 20 | 14 | 7
  Week 8: >=30% Reduction | 78 | 109 | 99 | 75
  Week 8: >=50% Reduction | 47 | 71 | 73 | 47
  Week 8: >=70% Reduction | 21 | 44 | 47 | 27
  Week 8: >=90% Reduction | 5 | 20 | 16 | 4
  Week 12: >=30% Reduction | 80 | 107 | 102 | 81
  Week 12: >=50% Reduction | 44 | 75 | 77 | 51
  Week 12: >=70% Reduction | 26 | 48 | 44 | 26
  Week 12: >=90% Reduction | 6 | 25 | 18 | 6
  Week 16: >=30% Reduction | 78 | 107 | 103 | 78
  Week 16: >=50% Reduction | 47 | 76 | 75 | 51
  Week 16: >=70% Reduction | 29 | 47 | 43 | 28
  Week 16: >=90% Reduction | 8 | 24 | 19 | 3

12. Secondary Outcome: Number of Participants With At Least (>=) 30 Percent (%), 50%, 70% and 90% Reduction From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Weeks 2, 4, 8, 12 and 16: mITT Population
Description: as for outcome 2
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 137 | 153 | 149 | 156
Participants
  Week 2: >=30% Reduction | 54 | 67 | 58 | 63
  Week 2: >=50% Reduction | 28 | 41 | 37 | 31
  Week 2: >=70% Reduction | 9 | 21 | 12 | 13
  Week 2: >=90% Reduction | 1 | 4 | 2 | 5
  Week 4: >=30% Reduction | 62 | 88 | 78 | 74
  Week 4: >=50% Reduction | 39 | 61 | 55 | 40
  Week 4: >=70% Reduction | 13 | 40 | 37 | 22
  Week 4: >=90% Reduction | 3 | 17 | 9 | 6
  Week 8: >=30% Reduction | 73 | 94 | 81 | 69
  Week 8: >=50% Reduction | 43 | 63 | 57 | 38
  Week 8: >=70% Reduction | 16 | 43 | 39 | 22
  Week 8: >=90% Reduction | 5 | 19 | 8 | 4
  Week 12: >=30% Reduction | 76 | 97 | 83 | 76
  Week 12: >=50% Reduction | 41 | 68 | 61 | 43
  Week 12: >=70% Reduction | 21 | 45 | 38 | 21
  Week 12: >=90% Reduction | 6 | 24 | 9 | 7
  Week 16: >=30% Reduction | 78 | 97 | 87 | 75
  Week 16: >=50% Reduction | 44 | 71 | 63 | 44
  Week 16: >=70% Reduction | 25 | 47 | 40 | 21
  Week 16: >=90% Reduction | 8 | 23 | 10 | 5

13. Secondary Outcome: Number of Participants With Cumulative Reduction From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 8: ITT Population
Description: The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to OA in the index joint (knee/hip) during the past 48 hours. It is calculated as the mean of the scores from the 5 individual questions scored on an NRS of 0 to 10, where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 to 10, where higher scores indicate higher pain. Participants with specified reduction (as percent) from baseline at Week 8 are reported.
Time Frame: Week 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
Participants
  Greater than (>) 0% Reduction | 121 | 149 | 134 | 139
  >=10% Reduction | 109 | 138 | 127 | 125
  >=20% Reduction | 91 | 125 | 110 | 101
  >=30% Reduction | 78 | 109 | 99 | 75
  >=40% Reduction | 54 | 93 | 86 | 57
  >=50% Reduction | 47 | 71 | 73 | 47
  >=60% Reduction | 31 | 62 | 61 | 38
  >=70% Reduction | 21 | 44 | 47 | 27
  >=80% Reduction | 11 | 30 | 28 | 10
  >=90% Reduction | 5 | 20 | 16 | 4
  100% Reduction | 0 | 12 | 5 | 2

14. Secondary Outcome: Number of Participants With Cumulative Reduction From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 8: mITT Population
Description: as for outcome 2
Time Frame: Week 8
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 137 | 153 | 149 | 156
Participants
  >0% Reduction | 108 | 127 | 115 | 119
  >=10% Reduction | 94 | 119 | 111 | 105
  >=20% Reduction | 83 | 106 | 92 | 92
  >=30% Reduction | 73 | 94 | 81 | 69
  >=40% Reduction | 51 | 80 | 67 | 51
  >=50% Reduction | 43 | 63 | 57 | 38
  >=60% Reduction | 29 | 54 | 47 | 31
  >=70% Reduction | 16 | 43 | 39 | 22
  >=80% Reduction | 14 | 26 | 22 | 11
  >=90% Reduction | 5 | 19 | 8 | 4
  100% Reduction | 1 | 11 | 3 | 1

15. Secondary Outcome: Number of Participants With Improvement of At Least (>=) 2 Points From Baseline in Patient Global Assessment (PGA) of Osteoarthritis at Weeks 2, 4, 8, 12 and 16: ITT Population
Description: as for outcome 7
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
Participants
  Week 2 | 16 | 24 | 19 | 17
  Week 4 | 17 | 45 | 37 | 19
  Week 8 | 13 | 36 | 42 | 17
  Week 12 | 17 | 40 | 47 | 23
  Week 16 | 18 | 38 | 44 | 18

16. Secondary Outcome: Number of Participants With Improvement of At Least (>=) 2 Points From Baseline in Patient Global Assessment (PGA) of Osteoarthritis at Weeks 2, 4, 8 12 and 16: mITT Population
Description: as for outcome 7
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 137 | 153 | 149 | 156
Participants
  Week 2 | 15 | 23 | 17 | 16
  Week 4 | 16 | 39 | 32 | 15
  Week 8 | 14 | 38 | 31 | 14
  Week 12 | 18 | 39 | 33 | 19
  Week 16 | 21 | 39 | 35 | 16

17. Secondary Outcome: Change From Baseline in Average Pain Score in the Index Knee or Index Hip at Weeks 1, 2, 3, 4, 6, 8, 10, 12, and 16: ITT Population
Description: Participants assessed daily average pain in the index joint (knee/hip) during the past 24 hours on an 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain). Higher score indicated greater pain. The baseline mean was calculated using the daily pain scores in the index joint (knee/hip) over the 3 days in the initial pain assessment period and the weekly mean was calculated using the daily pain scores in the index joint (knee/hip) within each assessment week.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 6, 8, 10, 12, and 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 138 | 160 | 148 | 155
units on a scale
  Baseline | 7.18 (1.80) | 7.28 (1.62) | 6.98 (1.84) | 7.03 (1.72)
  Change at Week 1 | -0.79 (1.30) | -1.71 (1.93) | -1.47 (1.84) | -1.15 (1.65)
  Change at Week 2 | -1.26 (1.63) | -1.96 (2.23) | -1.43 (2.13) | -1.54 (1.99)
  Change at Week 3 | -1.57 (1.73) | -2.27 (2.42) | -1.71 (2.29) | -1.67 (2.08)
  Change at Week 4 | -1.70 (1.81) | -2.65 (2.49) | -2.28 (2.60) | -1.76 (2.10)
  Change at Week 6 | -1.91 (1.95) | -2.87 (2.55) | -2.43 (2.66) | -1.94 (2.18)
  Change at Week 8 | -1.96 (1.99) | -2.82 (2.54) | -2.38 (2.72) | -1.83 (2.18)
  Change at Week 10 | -2.06 (2.16) | -2.92 (2.62) | -2.39 (2.72) | -1.89 (2.23)
  Change at Week 12 | -2.07 (2.27) | -2.94 (2.60) | -2.38 (2.67) | -1.88 (2.33)
  Change at Week 16 | -2.09 (2.31) | -2.90 (2.63) | -2.39 (2.68) | -1.86 (2.28)

18. Secondary Outcome: Change From Baseline in Average Pain Score in the Index Knee or Index Hip at Weeks 1, 2, 3, 4, 6, 8, 10, 12, and 16: mITT Population
Description: as for outcome 17
Time Frame: Baseline, Weeks 1, 2, 3, 4, 6, 8, 10, 12, and 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 134 | 152 | 147 | 153
units on a scale
  Baseline | 7.16 (1.81) | 7.31 (1.62) | 6.98 (1.84) | 7.05 (1.71)
  Change at Week 1 | -0.79 (1.24) | -1.71 (1.96) | -1.50 (1.81) | -1.16 (1.64)
  Change at Week 2 | -1.23 (1.59) | -1.99 (2.19) | -1.51 (2.10) | -1.46 (1.96)
  Change at Week 3 | -1.54 (1.74) | -2.28 (2.31) | -1.73 (2.20) | -1.58 (2.07)
  Change at Week 4 | -1.63 (1.85) | -2.70 (2.42) | -2.21 (2.52) | -1.70 (2.10)
  Change at Week 6 | -1.78 (1.96) | -2.92 (2.48) | -2.37 (2.58) | -1.85 (2.17)
  Change at Week 8 | -1.82 (2.00) | -2.88 (2.50) | -2.36 (2.63) | -1.78 (2.16)
  Change at Week 10 | -1.95 (2.17) | -2.98 (2.56) | -2.40 (2.63) | -1.83 (2.20)
  Change at Week 12 | -1.96 (2.27) | -3.00 (2.53) | -2.36 (2.61) | -1.83 (2.27)
  Change at Week 16 | -1.96 (2.31) | -2.97 (2.55) | -2.40 (2.63) | -1.84 (2.23)

19. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale Score at Weeks 2, 4, 8, 12, and 16: ITT Population
Description: The WOMAC stiffness subscale is a 2-item questionnaire used to assess the amount of stiffness experienced due to OA in the index joint (knee/hip) during past 48 hours. It is calculated as the mean of the scores from the 2 individual questions scored on NRS of 0 to 10; with higher scores indicating more stiffness. Total score range for WOMAC stiffness subscale score is 0 to 10, where higher scores indicate more stiffness. Stiffness is defined as a sensation of decreased ease in moving the index joint (knee/hip).
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
units on a scale
  Baseline | 7.22 (1.67) | 7.30 (1.92) | 7.15 (1.82) | 7.39 (1.72)
  Change at Week 2 | -1.49 (1.83) | -2.24 (2.50) | -2.19 (2.41) | -1.78 (2.16)
  Change at Week 4 | -1.88 (1.95) | -3.12 (2.70) | -3.08 (2.91) | -2.16 (2.35)
  Change at Week 8 | -1.92 (2.17) | -3.09 (2.60) | -3.28 (2.77) | -2.19 (2.43)
  Change at Week 12 | -2.15 (2.35) | -3.33 (2.75) | -3.31 (2.72) | -2.25 (2.45)
  Change at Week 16 | -2.20 (2.50) | -3.24 (2.73) | -3.25 (2.66) | -2.19 (2.40)

20. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale Score at Weeks 2, 4, 8, 12, and 16: mITT Population
Description: as for outcome 19
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 137 | 153 | 149 | 156
units on a scale
  Baseline | 7.22 (1.69) | 7.29 (1.93) | 7.16 (1.82) | 7.39 (1.72)
  Change at Week 2 | -1.38 (1.87) | -2.08 (2.53) | -1.90 (2.26) | -1.57 (2.13)
  Change at Week 4 | -1.71 (2.02) | -2.91 (2.82) | -2.61 (2.90) | -1.92 (2.36)
  Change at Week 8 | -1.77 (2.14) | -2.97 (2.74) | -2.72 (2.88) | -1.92 (2.34)
  Change at Week 12 | -2.01 (2.32) | -3.24 (2.88) | -2.77 (2.85) | -2.06 (2.40)
  Change at Week 16 | -2.14 (2.47) | -3.24 (2.83) | -2.83 (2.87) | -2.06 (2.37)

21. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Weeks 2, 4, 8, 12, and 16: ITT Population
Description: WOMAC: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain (5 items), stiffness (2 items) and physical function (17 items) in participants with OA of the index knee or index hip. WOMAC average score is the mean of WOMAC pain, physical function and stiffness subscale scores and ranges from 0 to 10, where higher score indicates worse response.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
units on a scale
  Baseline | 7.39 (1.32) | 7.48 (1.43) | 7.27 (1.40) | 7.50 (1.33)
  Change at Week 2 | -1.71 (1.67) | -2.29 (2.21) | -2.15 (2.04) | -1.94 (1.91)
  Change at Week 4 | -2.11 (1.88) | -3.24 (2.49) | -3.16 (2.58) | -2.38 (2.12)
  Change at Week 8 | -2.23 (2.05) | -3.32 (2.40) | -3.33 (2.49) | -2.35 (2.22)
  Change at Week 12 | -2.39 (2.20) | -3.49 (2.55) | -3.35 (2.45) | -2.41 (2.23)
  Change at Week 16 | -2.47 (2.33) | -3.42 (2.53) | -3.34 (2.39) | -2.39 (2.20)

22. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Weeks 2, 4, 8, 12, and 16: mITT Population
Description: as for outcome 21
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 137 | 153 | 149 | 156
units on a scale
  Baseline | 7.38 (1.34) | 7.50 (1.44) | 7.28 (1.40) | 7.51 (1.33)
  Change at Week 2 | -1.60 (1.70) | -2.14 (2.25) | -1.90 (1.96) | -1.74 (1.94)
  Change at Week 4 | -1.94 (1.93) | -2.99 (2.61) | -2.64 (2.61) | -2.08 (2.13)
  Change at Week 8 | -2.08 (2.03) | -3.13 (2.59) | -2.79 (2.60) | -2.07 (2.16)
  Change at Week 12 | -2.25 (2.19) | -3.34 (2.72) | -2.83 (2.60) | -2.20 (2.21)
  Change at Week 16 | -2.40 (2.36) | -3.36 (2.71) | -2.92 (2.62) | -2.20 (2.19)

23. Secondary Outcome: Change From Baseline in WOMAC Pain Subscale Item (Pain When Walking on a Flat Surface) at Weeks 2, 4, 8, 12, and 16: ITT Population
Description: Participants answered: "How much pain have you had when walking on a flat surface?" Participants responded by using a NRS of 0 to 10, where 0 = no pain and 10 = extreme pain. Higher score indicated greater pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
units on a scale
  Baseline | 7.58 (1.57) | 7.80 (1.45) | 7.67 (1.54) | 7.70 (1.66)
  Change at Week 2 | -2.01 (2.17) | -2.61 (2.53) | -2.43 (2.39) | -2.27 (2.17)
  Change at Week 4 | -2.46 (2.30) | -3.54 (2.72) | -3.58 (2.86) | -2.91 (2.42)
  Change at Week 8 | -2.70 (2.63) | -3.75 (2.64) | -3.82 (2.86) | -2.72 (2.50)
  Change at Week 12 | -2.85 (2.72) | -3.84 (2.80) | -3.85 (2.80) | -2.80 (2.58)
  Change at Week 16 | -2.91 (2.73) | -3.79 (2.75) | -3.76 (2.76) | -2.72 (2.48)

24. Secondary Outcome: Change From Baseline in WOMAC Pain Subscale Item (Pain When Walking on a Flat Surface) at Weeks 2, 4, 8, 12, and 16: mITT Population
Description: as for outcome 23
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 137 | 153 | 149 | 156
units on a scale
  Baseline | 7.60 (1.56) | 7.80 (1.46) | 7.68 (1.54) | 7.72 (1.62)
  Change at Week 2 | -1.85 (2.15) | -2.47 (2.55) | -2.19 (2.28) | -1.99 (2.15)
  Change at Week 4 | -2.26 (2.34) | -3.20 (2.73) | -2.98 (2.84) | -2.50 (2.37)
  Change at Week 8 | -2.50 (2.59) | -3.36 (2.77) | -3.19 (2.92) | -2.39 (2.33)
  Change at Week 12 | -2.66 (2.75) | -3.54 (2.92) | -3.23 (2.88) | -2.56 (2.44)
  Change at Week 16 | -2.83 (2.81) | -3.57 (2.90) | -3.32 (2.90) | -2.51 (2.37)

25. Secondary Outcome: Change From Baseline in WOMAC Pain Subscale Item (Pain When Going Up or Down Stairs) at Weeks 2, 4, 8, 12, and 16: ITT Population
Description: Participants answered: "How much pain have you had when going up or down stairs?" Participants responded by using a NRS of 0 to 10, where 0 = no pain and 10 = extreme pain. Higher score indicated greater pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
units on a scale
  Baseline | 8.59 (1.20) | 8.39 (1.29) | 8.45 (1.42) | 8.53 (1.37)
  Change at Week 2 | -2.06 (1.99) | -2.34 (2.45) | -2.39 (2.40) | -2.08 (2.10)
  Change at Week 4 | -2.64 (2.12) | -3.39 (2.78) | -3.48 (2.84) | -2.64 (2.31)
  Change at Week 8 | -2.77 (2.34) | -3.58 (2.81) | -3.74 (2.86) | -2.51 (2.37)
  Change at Week 12 | -2.87 (2.38) | -3.70 (2.98) | -3.76 (2.87) | -2.68 (2.48)
  Change at Week 16 | -3.02 (2.55) | -3.61 (2.86) | -3.75 (2.80) | -2.66 (2.45)

26. Secondary Outcome: Change From Baseline in WOMAC Pain Subscale Item (Pain When Going Up or Down Stairs) at Weeks 2, 4, 8, 12, and 16: mITT Population
Description: as for outcome 25
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 137 | 153 | 149 | 156
units on a scale
  Baseline | 8.59 (1.20) | 8.42 (1.27) | 8.44 (1.42) | 8.55 (1.35)
  Change at Week 2 | -1.90 (1.98) | -2.21 (2.45) | -2.06 (2.26) | -1.87 (2.16)
  Change at Week 4 | -2.44 (2.19) | -3.10 (2.82) | -2.81 (2.79) | -2.24 (2.28)
  Change at Week 8 | -2.62 (2.36) | -3.25 (2.86) | -3.04 (2.86) | -2.21 (2.29)
  Change at Week 12 | -2.71 (2.45) | -3.40 (2.99) | -3.11 (2.88) | -2.40 (2.44)
  Change at Week 16 | -2.91 (2.64) | -3.42 (2.92) | -3.24 (2.89) | -2.40 (2.42)

27. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36v2) Domain Scores at Week 12: ITT Population
Description: SF-36v2: standardized survey evaluating 8 health concepts (physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health). Total score for each health concept was scaled 0-100 (100 = highest level of functioning).
Time Frame: Baseline, Week 12
Population: ITT analysis set included all randomized participants who received at least 1 dose of randomized intravenous study medication (either tanezumab or placebo). Missing data were imputed using baseline observation carried forward (BOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
units on a scale
  General Health: Baseline | 55.28 (22.21) | 58.35 (19.26) | 60.01 (21.71) | 55.47 (18.53)
  General Health: Change at Week 12 | 1.89 (10.11) | 2.22 (9.37) | 2.85 (10.47) | 1.21 (10.66)
  Physical Function: Baseline | 29.09 (18.40) | 31.80 (19.15) | 32.14 (18.61) | 28.55 (17.70)
  Physical Function: Change at Week 12 | 6.03 (15.83) | 10.88 (21.94) | 5.57 (15.15) | 4.05 (13.30)
  Role Physical: Baseline | 37.81 (22.80) | 40.72 (24.20) | 39.46 (21.74) | 36.75 (21.53)
  Role Physical: Change at Week 12 | 7.14 (17.54) | 10.83 (22.26) | 6.17 (16.53) | 5.62 (18.36)
  Bodily Pain: Baseline | 28.43 (13.80) | 28.80 (14.51) | 29.08 (15.48) | 27.23 (14.15)
  Bodily Pain: Change at Week 12 | 6.38 (15.63) | 12.38 (21.23) | 8.32 (16.82) | 6.36 (13.92)
  Vitality: Baseline | 46.37 (20.06) | 48.95 (20.59) | 47.25 (21.03) | 45.33 (20.61)
  Vitality: Change at Week 12 | 3.10 (10.58) | 4.19 (12.99) | 3.08 (12.33) | 2.25 (13.99)
  Social Function: Baseline | 57.36 (26.18) | 62.34 (27.42) | 61.58 (26.63) | 57.91 (25.84)
  Social Function: Change at Week 12 | 5.41 (15.69) | 5.28 (16.40) | 4.50 (17.46) | 4.11 (17.07)
  Role Emotional: Baseline | 60.22 (31.11) | 64.70 (31.38) | 63.89 (30.48) | 60.81 (30.92)
  Role Emotional: Change at Week 12 | 3.72 (16.01) | 4.92 (19.58) | 2.06 (19.09) | 0.42 (15.19)
  Mental Health: Baseline | 68.40 (20.39) | 69.13 (19.60) | 68.27 (20.37) | 67.59 (19.26)
  Mental Health: Change at Week 12 | 1.03 (9.77) | 1.37 (10.61) | 2.20 (10.61) | 0.70 (12.00)

28. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36v2) Domain Scores at Week 12: mITT Population
Description: as for outcome 27
Time Frame: Baseline, Week 12
Population: mITT analysis set included all participants in ITT analysis set who had Week 8 visit on or before 23 June 2010 (effective date of the US FDA imposed clinical hold). Missing data were imputed using BOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 137 | 153 | 149 | 156
units on a scale
  General Health: Baseline | 55.61 (22.01) | 59.08 (18.43) | 60.21 (21.64) | 55.56 (18.60)
  General Health: Change at Week 12 | 1.85 (9.14) | 1.39 (8.49) | 2.61 (9.00) | 0.74 (8.71)
  Physical Function: Baseline | 29.18 (18.62) | 31.54 (19.35) | 32.29 (18.59) | 28.50 (17.75)
  Physical Function: Change at Week 12 | 5.36 (15.35) | 8.84 (19.48) | 3.76 (13.07) | 2.82 (11.81)
  Role Physical: Baseline | 37.73 (23.09) | 41.30 (24.44) | 39.43 (21.81) | 36.66 (21.07)
  Role Physical: Change at Week 12 | 6.07 (16.27) | 9.60 (20.20) | 5.49 (15.56) | 4.21 (15.61)
  Bodily Pain: Baseline | 28.55 (13.96) | 29.06 (14.52) | 29.21 (15.45) | 27.18 (14.06)
  Bodily Pain: Change at Week 12 | 5.54 (14.93) | 10.53 (20.14) | 7.41 (16.12) | 5.14 (12.93)
  Vitality: Baseline | 46.30 (20.23) | 48.73 (20.58) | 47.32 (21.09) | 45.11 (20.54)
  Vitality: Change at Week 12 | 2.97 (10.14) | 4.33 (12.61) | 3.02 (11.22) | 1.64 (12.40)
  Social Function: Baseline | 57.39 (26.15) | 62.58 (27.64) | 61.66 (26.70) | 57.93 (25.76)
  Social Function: Change at Week 12 | 4.65 (15.08) | 5.07 (15.47) | 5.12 (16.38) | 3.29 (15.43)
  Role Emotional: Baseline | 60.04 (31.35) | 64.54 (31.10) | 63.93 (30.58) | 60.68 (30.92)
  Role Emotional: Change at Week 12 | 3.89 (14.92) | 4.52 (19.19) | 2.07 (17.00) | -0.11 (11.86)
  Mental Health: Baseline | 68.03 (20.53) | 69.22 (19.57) | 68.36 (20.41) | 67.53 (19.36)
  Mental Health: Change at Week 12 | 0.62 (9.44) | 1.70 (9.82) | 2.55 (9.09) | 0.48 (10.06)

29. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36v2) Physical and Mental Component Aggregate Scores at Week 12: ITT Population
Description: SF-36v2: standardized survey evaluating 8 health concepts (physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health). Total score for each health concept was scaled 0-100 (100=highest level of functioning). For obtaining physical and mental component scores, z-score for each scale = (observed score - mean score for general 1990 United States [US] population)/corresponding standard deviation. The 2 component scores were obtained by multiplying each aspect z-score by physical or mental factor score coefficient (1990 general US population) and summing the eight products. Component scores indicated how many standard deviations higher (in case of positive z-score [better functioning])/lower (in case of negative z-score [worse functioning]) participant's value was relative to the mean of the reference population. Change from baseline >0 indicates an improvement.
Time Frame: Baseline, Week 12
Population: ITT analysis set included all randomized participants who received at least 1 dose of randomized intravenous study medication (either tanezumab or placebo). Missing data were imputed using BOCF.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
z-score
  Mental Component Aggregate: Baseline | -0.28 (1.27) | -0.13 (1.27) | -0.20 (1.28) | -0.28 (1.27)
  Mental Component Aggregate: Change at Week 12 | 0.08 (0.53) | 0.04 (0.65) | 0.07 (0.72) | 0.01 (0.67)
  Physical Component Aggregate: Baseline | -1.99 (0.72) | -1.91 (0.64) | -1.88 (0.69) | -2.03 (0.64)
  Physical Component Aggregate: Change at Week 12 | 0.26 (0.63) | 0.47 (0.88) | 0.28 (0.57) | 0.23 (0.57)

30. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36v2) Physical and Mental Component Aggregate Scores at Week 12: mITT Population
Description: as for outcome 29
Time Frame: Baseline, Week 12
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 137 | 153 | 149 | 156
z-score
  Mental Component Aggregate: Baseline | -0.30 (1.27) | -0.13 (1.26) | -0.19 (1.28) | -0.29 (1.27)
  Mental Component Aggregate: Change at Week 12 | 0.08 (0.51) | 0.07 (0.61) | 0.11 (0.64) | -0.00 (0.56)
  Physical Component Aggregate: Baseline | -1.98 (0.72) | -1.90 (0.65) | -1.88 (0.69) | -2.03 (0.63)
  Physical Component Aggregate: Change at Week 12 | 0.23 (0.60) | 0.38 (0.78) | 0.22 (0.53) | 0.18 (0.51)

31. Secondary Outcome: Change From Baseline in Euro Quality of Life-5 Dimension (EQ-5D) - Health State Profile Utility Score at Week 12: ITT Population
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains/items: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. Each item has 3 possible responses: no problems (level 1), some problems (level 2), and extreme problems (level 3). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Week 12
Population: ITT analysis set. Here 'overall number of participants analyzed' signifies participants who were evaluable for this measure and 'number analyzed' signifies participants who were evaluable at specified time-point for each treatment arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 140 | 161 | 150 | 156
units on a scale
  Baseline | 0.39 (0.31) | 0.41 (0.31) | 0.43 (0.29) | 0.38 (0.30)
  Change at Week 12: number analyzed (Participants) | 56 | 61 | 57 | 59
  Change at Week 12 | 0.25 (0.36) | 0.33 (0.34) | 0.22 (0.31) | 0.14 (0.28)

32. Secondary Outcome: Change From Baseline in Euro Quality of Life-5 Dimension (EQ-5D) - Health State Profile Utility Score at Week 12: mITT Population
Description: as for outcome 31
Time Frame: Baseline, Week 12
Population: mITT analysis set. Here 'overall number of participants analyzed' signifies participants who were evaluable for this measure and 'number analyzed' signifies participants who were evaluable at specified time-point for each treatment arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 136 | 153 | 149 | 154
units on a scale
  Baseline | 0.40 (0.31) | 0.41 (0.31) | 0.43 (0.30) | 0.38 (0.30)
  Change at Week 12: number analyzed (Participants) | 56 | 61 | 57 | 59
  Change at Week 12 | 0.25 (0.36) | 0.33 (0.34) | 0.22 (0.31) | 0.14 (0.28)

33. Secondary Outcome: Number of Participants With Change From Baseline in Euro Quality of Life-5 Dimension (EQ-5D) - Individual Dimensions at Week 12: ITT Population
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 dimensions/domains/items: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. Each item has 3 possible responses: no dysfunction (level 1), moderate/some dysfunction (level 2), and extreme dysfunction (level 3). Change from baseline at Week 12 is defined as: Improved (positive change), No change, and Worsened (negative change). Number of participants with response is reported.
Time Frame: Baseline, Week 12
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 140 | 161 | 150 | 156
Participants
  Mobility, Baseline: Level 1 | 8 | 15 | 10 | 7
  Mobility, Baseline: Level 2 | 132 | 146 | 140 | 148
  Mobility, Baseline: Level 3 | 0 | 0 | 0 | 1
  Mobility, Change at Wk 12: Improved: number analyzed (Participants) | 56 | 61 | 57 | 59
  Mobility, Change at Wk 12: Improved | 12 | 29 | 17 | 4
  Mobility, Change at Wk 12: No Change: number analyzed (Participants) | 56 | 61 | 57 | 59
  Mobility, Change at Wk 12: No Change | 43 | 31 | 39 | 53
  Mobility, Change at Wk 12: Worsened: number analyzed (Participants) | 56 | 61 | 57 | 59
  Mobility, Change at Wk 12: Worsened | 1 | 1 | 1 | 2
  Self-care, Baseline: Level 1 | 93 | 122 | 99 | 108
  Self-care, Baseline: Level 2 | 45 | 38 | 50 | 48
  Self-care, Baseline: Level 3 | 2 | 1 | 1 | 0
  Self-care, Change at Week 12: Improved: number analyzed (Participants) | 56 | 61 | 57 | 59
  Self-care, Change at Week 12: Improved | 15 | 12 | 17 | 10
  Self-care, Change at Week 12: No Change: number analyzed (Participants) | 56 | 61 | 57 | 59
  Self-care, Change at Week 12: No Change | 39 | 46 | 38 | 44
  Self-care, Change at Week 12: Worsened: number analyzed (Participants) | 56 | 61 | 57 | 59
  Self-care, Change at Week 12: Worsened | 2 | 3 | 2 | 5
  Usual Activities, Baseline: Level 1 | 15 | 21 | 19 | 15
  Usual Activities, Baseline: Level 2 | 123 | 134 | 125 | 136
  Usual Activities, Baseline: Level 3 | 2 | 6 | 6 | 5
  Usual Activities, Change at Week 12: Improved: number analyzed (Participants) | 56 | 61 | 57 | 59
  Usual Activities, Change at Week 12: Improved | 15 | 27 | 15 | 21
  Usual Activities, Change at Week 12: No Change: number analyzed (Participants) | 56 | 61 | 57 | 59
  Usual Activities, Change at Week 12: No Change | 36 | 32 | 41 | 36
  Usual Activities, Change at Week 12: Worsened: number analyzed (Participants) | 56 | 61 | 57 | 59
  Usual Activities, Change at Week 12: Worsened | 5 | 2 | 1 | 2
  Pain and Discomfort, Baseline: Level 1: number analyzed (Participants) | 139 | 161 | 149 | 156
  Pain and Discomfort, Baseline: Level 1 | 2 | 1 | 0 | 1
  Pain and Discomfort, Baseline: Level 2: number analyzed (Participants) | 139 | 161 | 149 | 156
  Pain and Discomfort, Baseline: Level 2 | 77 | 92 | 94 | 83
  Pain and Discomfort, Baseline: Level 3: number analyzed (Participants) | 139 | 161 | 149 | 156
  Pain and Discomfort, Baseline: Level 3 | 60 | 68 | 55 | 72
  Pain and Discomfort, Change at Week 12: Improved: number analyzed (Participants) | 55 | 61 | 57 | 59
  Pain and Discomfort, Change at Week 12: Improved | 23 | 32 | 21 | 17
  Pain and Discomfort, Change at Week 12: No Change: number analyzed (Participants) | 55 | 61 | 57 | 59
  Pain and Discomfort, Change at Week 12: No Change | 29 | 28 | 35 | 39
  Pain and Discomfort, Change at Week 12: Worsened: number analyzed (Participants) | 55 | 61 | 57 | 59
  Pain and Discomfort, Change at Week 12: Worsened | 3 | 1 | 1 | 3
  Anxiety and Depression, Baseline: Level 1: number analyzed (Participants) | 140 | 161 | 149 | 156
  Anxiety and Depression, Baseline: Level 1 | 79 | 86 | 92 | 84
  Anxiety and Depression, Baseline: Level 2: number analyzed (Participants) | 140 | 161 | 149 | 156
  Anxiety and Depression, Baseline: Level 2 | 52 | 68 | 52 | 68
  Anxiety and Depression, Baseline: Level 3: number analyzed (Participants) | 140 | 161 | 149 | 156
  Anxiety and Depression, Baseline: Level 3 | 9 | 7 | 5 | 4
  Anxiety and Depression, Change at Week 12: Improved: number analyzed (Participants) | 56 | 61 | 57 | 59
  Anxiety and Depression, Change at Week 12: Improved | 16 | 16 | 12 | 9
  Anxiety and Depression, Change at Week 12: No Change: number analyzed (Participants) | 56 | 61 | 57 | 59
  Anxiety and Depression, Change at Week 12: No Change | 35 | 40 | 37 | 42
  Anxiety and Depression, Change at Week 12: Worsened: number analyzed (Participants) | 56 | 61 | 57 | 59
  Anxiety and Depression, Change at Week 12: Worsened | 5 | 5 | 8 | 8

34. Secondary Outcome: Number of Participants With Change From Baseline in Euro Quality of Life-5 Dimension (EQ-5D) - Individual Dimensions at Week 12: mITT Population
Description: as for outcome 33
Time Frame: Baseline, Week 12
Population: mITT analysis set. Here 'overall number of participants analyzed' signifies participants who were evaluable for this measure and 'number anlayzed' signifies participants who were evaluable at specified time-point for each treatment arm, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 136 | 153 | 149 | 154
Participants
  Mobility, Baseline: Level 1 | 8 | 14 | 10 | 7
  Mobility, Baseline: Level 2 | 128 | 139 | 139 | 146
  Mobility, Baseline: Level 3 | 0 | 0 | 0 | 1
  Mobility, Change at Week 12: Improved: number analyzed (Participants) | 56 | 61 | 57 | 59
  Mobility, Change at Week 12: Improved | 12 | 29 | 17 | 4
  Mobility, Change at Week 12: No Change: number analyzed (Participants) | 56 | 61 | 57 | 59
  Mobility, Change at Week 12: No Change | 43 | 31 | 39 | 53
  Mobility, Change at Week 12: Worsened: number analyzed (Participants) | 56 | 61 | 57 | 59
  Mobility, Change at Week 12: Worsened | 1 | 1 | 1 | 2
  SC, Baseline: Level 1 | 91 | 118 | 99 | 108
  Self-care, Baseline: Level 2 | 43 | 34 | 49 | 46
  Self-care, Baseline: Level 3 | 2 | 1 | 1 | 0
  Self-care, Change at Week 12: Improved: number analyzed (Participants) | 56 | 61 | 57 | 59
  Self-care, Change at Week 12: Improved | 15 | 12 | 17 | 10
  Self-care, Change at Week 12: No Change: number analyzed (Participants) | 56 | 61 | 57 | 59
  Self-care, Change at Week 12: No Change | 39 | 46 | 38 | 44
  Self-care, Change at Week 12: Worsened: number analyzed (Participants) | 56 | 61 | 57 | 59
  Self-care, Change at Week 12: Worsened | 2 | 3 | 2 | 5
  Usual Activities, Baseline: Level 1 | 15 | 20 | 19 | 15
  Usual Activities, Baseline: Level 2 | 119 | 128 | 124 | 134
  Usual Activities, Baseline: Level 3 | 2 | 5 | 6 | 5
  Usual Activities, Change at Week 12: Improved: number analyzed (Participants) | 56 | 61 | 57 | 59
  Usual Activities, Change at Week 12: Improved | 15 | 27 | 15 | 21
  Usual Activities, Change at Week 12: No Change: number analyzed (Participants) | 56 | 61 | 57 | 59
  Usual Activities, Change at Week 12: No Change | 36 | 32 | 41 | 36
  Usual Activities, Change at Week 12: Worsened: number analyzed (Participants) | 56 | 61 | 57 | 59
  Usual Activities, Change at Week 12: Worsened | 5 | 2 | 1 | 2
  Pain and Discomfort, Baseline: Level 1: number analyzed (Participants) | 135 | 153 | 148 | 154
  Pain and Discomfort, Baseline: Level 1 | 2 | 1 | 0 | 1
  Pain and Discomfort, Baseline: Level 2: number analyzed (Participants) | 135 | 153 | 148 | 154
  Pain and Discomfort, Baseline: Level 2 | 77 | 87 | 93 | 82
  Pain and Discomfort, Baseline: Level 3: number analyzed (Participants) | 135 | 153 | 148 | 154
  Pain and Discomfort, Baseline: Level 3 | 56 | 65 | 55 | 71
  Pain and Discomfort, Change at Week 12: Improved: number analyzed (Participants) | 55 | 61 | 57 | 59
  Pain and Discomfort, Change at Week 12: Improved | 23 | 32 | 21 | 17
  Pain and Discomfort, Change at Week 12: No Change: number analyzed (Participants) | 55 | 61 | 57 | 59
  Pain and Discomfort, Change at Week 12: No Change | 29 | 28 | 35 | 39
  Pain and Discomfort, Change at Week 12: Worsened: number analyzed (Participants) | 55 | 61 | 57 | 59
  Pain and Discomfort, Change at Week 12: Worsened | 3 | 1 | 1 | 3
  Anxiety and Depression, Baseline: Level 1: number analyzed (Participants) | 136 | 153 | 148 | 154
  Anxiety and Depression, Baseline: Level 1 | 76 | 82 | 92 | 83
  Anxiety and Depression, Baseline: Level 2: number analyzed (Participants) | 136 | 153 | 148 | 154
  Anxiety and Depression, Baseline: Level 2 | 51 | 64 | 51 | 67
  Anxiety and Depression, Baseline: Level 3: number analyzed (Participants) | 136 | 153 | 148 | 154
  Anxiety and Depression, Baseline: Level 3 | 9 | 7 | 5 | 4
  Anxiety and Depression, Change at Week 12: Improved: number analyzed (Participants) | 56 | 61 | 57 | 59
  Anxiety and Depression, Change at Week 12: Improved | 16 | 16 | 12 | 9
  Anxiety and Depression, Change at Week 12: No Change: number analyzed (Participants) | 56 | 61 | 57 | 59
  Anxiety and Depression, Change at Week 12: No Change | 35 | 40 | 37 | 42
  Anxiety and Depression, Change at Week 12: Worsened: number analyzed (Participants) | 56 | 61 | 57 | 59
  Anxiety and Depression, Change at Week 12: Worsened | 5 | 5 | 8 | 8

35. Secondary Outcome: Number of Participants Who Discontinued From Study Due to Lack of Efficacy
Time Frame: Baseline up to Week 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of randomized intravenous study medication (either tanezumab or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
Participants | 10 | 6 | 5 | 12

36. Secondary Outcome: Time to Discontinuation From Study Due to Lack of Efficacy
Time Frame: Baseline up to Week 24
Population: Analysis set included participants from ITT analysis set who discontinued study due to lack of efficacy.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 10 | 6 | 5 | 12
days | 29.0 [8 to 182] | 43.0 [15 to 84] | 56.0 [22 to 106] | 30.0 [11 to 152]

37. Secondary Outcome: Number of Participants With Rescue Medication (RM) Usage
Description: In the event of inadequate pain relief for OA during the double-blind treatment period, participants were allowed to take up to 3000 mg of acetaminophen (tablet/capsule/caplets) per day up to 3 days per week as a rescue medication.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
Participants
  Week 2: number analyzed (Participants) | 128 | 144 | 142 | 150
  Week 2 | 90 | 85 | 99 | 90
  Week 4: number analyzed (Participants) | 131 | 146 | 144 | 150
  Week 4 | 76 | 65 | 79 | 85
  Week 8: number analyzed (Participants) | 131 | 147 | 144 | 151
  Week 8 | 67 | 63 | 65 | 77
  Week 12: number analyzed (Participants) | 131 | 147 | 144 | 151
  Week 12 | 68 | 52 | 61 | 78
  Week 16: number analyzed (Participants) | 132 | 147 | 144 | 151
  Week 16 | 68 | 50 | 59 | 72

38. Secondary Outcome: Number of Days With Rescue Medication (RM) Usage
Description: In the event of inadequate pain relief for OA during the double-blind treatment period, participants were allowed to take up to 3000 mg of acetaminophen (tablet/capsule/caplets) per day up to 3 days per week as a rescue medication. Results are shown in number of days of rescue medication usage per week.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: ITT analysis set. Missing data were imputed using LOCF. Here 'overall number of participants analyzed' signifies participants who were evaluable for this measure and 'number analyzed' signifies participants who were evaluable at specified time-point for each treatment arm, respectively.
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 132 | 147 | 144 | 151
days per week
  Week 2: number analyzed (Participants) | 128 | 144 | 142 | 150
  Week 2 | 2.72 (2.66) | 2.03 (2.46) | 2.58 (2.58) | 2.35 (2.69)
  Week 4: number analyzed (Participants) | 131 | 146 | 144 | 150
  Week 4 | 2.40 (2.72) | 1.60 (2.43) | 1.95 (2.51) | 2.27 (2.68)
  Week 8: number analyzed (Participants) | 131 | 147 | 144 | 151
  Week 8 | 2.11 (2.65) | 1.33 (2.24) | 1.72 (2.52) | 1.75 (2.38)
  Week 12: number analyzed (Participants) | 131 | 147 | 144 | 151
  Week 12 | 1.82 (2.39) | 1.20 (2.24) | 1.63 (2.41) | 1.74 (2.37)
  Week 16 | 1.73 (2.30) | 1.02 (1.99) | 1.40 (2.25) | 1.67 (2.39)

39. Secondary Outcome: Amount of Rescue Medication Used
Description: In the event of inadequate pain relief for OA during the double-blind treatment period, participants were allowed to take up to 3000 mg of acetaminophen (tablet/capsule/caplets) per day up to 3 days per week as a rescue medication. Results are presented as total dose of acetaminophen (in mg) per week.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: mg per week
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 132 | 147 | 144 | 151
mg per week
  Week 2: number analyzed (Participants) | 128 | 144 | 142 | 150
  Week 2 | 4109.38 (5190.82) | 2684.03 (4193.21) | 3510.56 (4321.51) | 3553.33 (5395.79)
  Week 4: number analyzed (Participants) | 131 | 146 | 144 | 150
  Week 4 | 3293.89 (4412.77) | 2136.99 (3741.44) | 2614.58 (4221.46) | 3373.33 (4886.01)
  Week 8: number analyzed (Participants) | 131 | 147 | 144 | 151
  Week 8 | 3000.00 (4277.85) | 1659.86 (3092.18) | 2336.81 (4033.87) | 2539.74 (4653.86)
  Week 12: number analyzed (Participants) | 131 | 147 | 144 | 151
  Week 12 | 2561.07 (3651.14) | 1394.56 (2893.80) | 2333.33 (4189.56) | 2360.93 (3786.45)
  Week 16 | 2412.88 (3416.67) | 1159.86 (2619.07) | 1965.28 (3865.60) | 2420.53 (4121.12)

40. Secondary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Weeks 2, 4, 8, 12, 16, and 18
Description: NIS: 74 items, assess muscle weakness, reflexes and sensation; scored separately for left, right limbs (37 items for each side). Components of muscle weakness are 24 items and scored on scale 0 (normal) to 4 (paralysis), higher score=greater weakness. Components of reflexes and sensation are 13 items and scored 0 = normal, 1= decreased, or 2 = absent. Total NIS score is the sum of the left and right limb scores. Total possible NIS score range 0 to 244, higher score=greater impairment.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, and 18
Population: ITT analysis set. Missing data were imputed using LOCF. Here 'number analyzed' signifies participants who were evaluable at specified time-point for each treatment arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
units on a scale
  Baseline | 1.43 (4.93) | 1.01 (3.11) | 1.32 (5.83) | 1.73 (4.10)
  Change at Week 2: number analyzed (Participants) | 133 | 151 | 141 | 152
  Change at Week 2 | -0.42 (3.04) | -0.22 (1.40) | -0.13 (0.79) | -0.16 (1.09)
  Change at Week 4: number analyzed (Participants) | 137 | 157 | 145 | 156
  Change at Week 4 | -0.09 (1.45) | -0.33 (2.00) | -0.28 (1.68) | -0.31 (1.59)
  Change at Week 8: number analyzed (Participants) | 139 | 157 | 149 | 156
  Change at Week 8 | -0.18 (1.93) | -0.22 (2.07) | -0.22 (1.51) | -0.39 (2.32)
  Change at Week 12: number analyzed (Participants) | 139 | 157 | 149 | 156
  Change at Week 12 | -0.19 (1.29) | -0.13 (4.13) | -0.33 (1.81) | -0.33 (1.79)
  Change at Week 16: number analyzed (Participants) | 139 | 158 | 149 | 156
  Change at Week 16 | -0.40 (1.94) | -0.14 (3.78) | -0.28 (1.74) | -0.53 (2.38)
  Change at Week 18: number analyzed (Participants) | 139 | 158 | 149 | 156
  Change at Week 18 | -0.25 (1.25) | -0.02 (2.91) | -0.25 (1.64) | -0.18 (2.13)

41. Secondary Outcome: Number of Participants With Anti-Drug (Tanezumab) Antibody (ADA)
Description: Human serum samples were analyzed for the presence or absence of anti-tanezumab antibodies by using the semi-quantitative enzyme-linked immunosorbent assay (ELISA). Only participants receiving tanezumab were to be analyzed for this measure. A participant may be represented in more than 1 category.
Time Frame: Baseline, Week 8 and 18
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 156 | 144
Participants
  Baseline | 0 | 1
  Week 8: number analyzed (Participants) | 124 | 107
  Week 8 | 1 | 2
  Week 18: number analyzed (Participants) | 117 | 109
  Week 18 | 0 | 0

42. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 112 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included SAEs as well as non-serious AEs which occurred during the trial.
Time Frame: Baseline up to 112 days after last intravenous dose
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
Participants
  AEs | 50 | 72 | 61 | 100
  SAEs | 2 | 4 | 3 | 4

43. Secondary Outcome: Number of Participants With Pre-Specified Opioid-Related Adverse Events According to Severity
Description: Pre-specified opioid-related adverse events: fatigue, drowsiness, inability to concentrate, nausea, dizziness, constipation, itching, difficulty urinating, confusion and vomiting. Number of participants who experienced any of the pre-specified opioid-related adverse event are reported. Pre-specified opioid-related adverse events were assessed according to severity: mild (did not interfere with participant's usual function); moderate (interfered to some extent with participant's usual function); and severe (interfered significantly with participant's usual function).
Time Frame: Baseline up to 112 days after last intravenous dose
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
Participants
  Fatigue: Mild | 0 | 2 | 1 | 6
  Fatigue: Moderate | 1 | 0 | 0 | 1
  Nausea: Mild | 0 | 5 | 3 | 14
  Nausea: Moderate | 0 | 1 | 0 | 11
  Dizziness: Mild | 2 | 2 | 3 | 10
  Constipation: Mild | 1 | 1 | 1 | 16
  Constipation: Moderate | 1 | 1 | 0 | 8
  Vomiting: Mild | 1 | 0 | 0 | 10
  Vomiting: Moderate | 0 | 1 | 0 | 5

44. Secondary Outcome: Number of Participants With Adverse Event of Abnormal Peripheral Sensation According to Severity
Description: Adverse event of abnormal peripheral sensation: allodynia, burning sensation, decreased vibratory sense, dysaesthesia, hyperaesthesia, hyperpathia, hypoaesthesia, neuralgia, neuritis, neuropathy peripheral, pallanesthesia, paraesthesia, paraesthesia oral, peripheral sensory neuropathy, polyneuropathy, sensory disturbance, sensory loss and thermohypoaesthesia. Adverse event of abnormal peripheral sensation was assessed according to severity: mild (did not interfere with participant's usual function); moderate (interfered to some extent with participant's usual function); and severe (interfered significantly with participant's usual function).
Time Frame: Baseline up to 112 days after last intravenous dose
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
Participants
  Burning Sensation: Mild | 0 | 0 | 1 | 0
  Decreased Vibratory Sense: Mild | 0 | 1 | 2 | 0
  Dysaesthesia: Mild | 1 | 0 | 0 | 1
  Hyperaesthesia: Mild | 0 | 0 | 2 | 0
  Hyperaesthesia: Moderate | 0 | 1 | 0 | 0
  Hypoaesthesia: Mild | 0 | 1 | 3 | 2
  Hypoaesthesia: Moderate | 0 | 2 | 0 | 0
  Hypoaesthesia: Severe | 0 | 1 | 0 | 0
  Neuropathy peripheral: Moderate | 0 | 1 | 0 | 0
  Paraesthesia: Mild | 0 | 4 | 3 | 1
  Paraesthesia: Moderate | 1 | 2 | 0 | 0

45. Secondary Outcome: Tanezumab Plasma Concentration
Description: Plasma concentration of tanezumab was measured using a validated, sensitive and specific enzyme-linked immunosorbent assay (ELISA). Only participants receiving tanezumab were to be analyzed for this measure.
Time Frame: Predose, 1 hour post-dose on Day 1, Week 8; Week 18
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 157 | 145
nanogram per milliliter (ng/mL)
  Predose, Day 1 | 36.96 (160.10) | 124.1 (601.80)
  1 hour post-dose, Day 1: number analyzed (Participants) | 121 | 111
  1 hour post-dose, Day 1 | 4192 (11266) | 5690 (10616)
  Predose, Week 8: number analyzed (Participants) | 122 | 108
  Predose, Week 8 | 207.0 (288.96) | 402.6 (257.29)
  1 hour post-dose, Week 8: number analyzed (Participants) | 64 | 53
  1 hour post-dose, Week 8 | 2259 (2349.1) | 3583 (1754.7)
  Week 18: number analyzed (Participants) | 113 | 110
  Week 18 | 87.05 (135.30) | 240.2 (386.98)

46. Secondary Outcome: Total Nerve Growth Factor (NGF) Serum Concentration
Description: Serum samples were analyzed for determining total NGF concentration. Total NGF was analyzed using a validated, sensitive, and specific immune-affinity enrichment liquid chromatography tandem mass spectrometric (IA/LC/MS/MS) method.
Time Frame: Predose, 1 hour post-dose on Day 1, Week 8; Predose: Week 18
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 116 | 128 | 124 | 119
picogram per milliliter (pg/mL)
  Predose, Day 1 | 58.1 (205.1) | 89.3 (538.1) | 138.2 (770.7) | 38.5 (10.8)
  1 hour post-dose, Day 1: number analyzed (Participants) | 101 | 123 | 111 | 114
  1 hour post-dose, Day 1 | 55.8 (172.9) | 133.9 (483.5) | 163.8 (565.2) | 39.0 (16.7)
  Predose, Week 8: number analyzed (Participants) | 76 | 123 | 106 | 87
  Predose, Week 8 | 92.6 (384.2) | 2152.2 (1040.8) | 3160.6 (1183.4) | 45.5 (13.2)
  1 hour post-dose, Week 8: number analyzed (Participants) | 47 | 70 | 64 | 43
  1 hour post-dose, Week 8 | 39.8 (9.9) | 2181.2 (1070.5) | 3026.0 (976.1) | 44.0 (22.0)
  Predose, Week 18: number analyzed (Participants) | 83 | 113 | 110 | 87
  Predose, Week 18 | 41.0 (15.2) | 1437.1 (1296.0) | 2365.4 (1402.4) | 48.7 (25.3)

47. Other Pre Specified Outcome: Number of Participants With Intravenous (IV) Doses of Study Medication
Description: Number of participants are reported based on the maximum number of IV doses of either tanezumab or placebo received.
Time Frame: Day 1 up to Week 16
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Number analyzed (Participants) | 141 | 161 | 150 | 158
Participants
  Number of IV Doses: 1 | 79 | 89 | 85 | 97
  Number of IV Doses: 2 | 62 | 72 | 65 | 61

ADVERSE EVENTS:
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study.
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Oxycodone CR
Serious Adverse Events (participants affected / at risk) | 2/141 | 4/161 | 3/150 | 4/158
Other Adverse Events (participants affected / at risk) | 36/141 | 43/161 | 33/150 | 82/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=141) | Tanezumab 5 mg (N=161) | Tanezumab 10 mg (N=150) | Oxycodone CR (N=158)
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 0
Drug ineffective (General disorders) | 1 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Clostridial infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia primary atypical (Infections and infestations) | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=141) | Tanezumab 5 mg (N=161) | Tanezumab 10 mg (N=150) | Oxycodone CR (N=158)
Constipation (Gastrointestinal disorders) | 2 | 2 | 1 | 24
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 3 | 1
Nausea (Gastrointestinal disorders) | 0 | 6 | 3 | 25
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 15
Fatigue (General disorders) | 1 | 2 | 1 | 7
Oedema peripheral (General disorders) | 3 | 4 | 4 | 3
Bronchitis (Infections and infestations) | 1 | 4 | 1 | 2
Nasopharyngitis (Infections and infestations) | 6 | 3 | 4 | 3
Urinary tract infection (Infections and infestations) | 4 | 4 | 2 | 4
Fall (Injury, poisoning and procedural complications) | 3 | 4 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 8 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 4 | 3
Dizziness (Nervous system disorders) | 2 | 2 | 3 | 10
Headache (Nervous system disorders) | 7 | 5 | 5 | 8
Hypoaesthesia (Nervous system disorders) | 0 | 4 | 3 | 2
Paraesthesia (Nervous system disorders) | 1 | 6 | 3 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 7
Insomnia (Psychiatric disorders) | 1 | 0 | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 10
Hypertension (Vascular disorders) | 2 | 2 | 1 | 5

LIMITATIONS AND CAVEATS:
Due to the US FDA imposed clinical hold (effective 23 June 2010), study was terminated early and planned sample size was not reached. The primary time-point was changed from Week 16 to Week 8, as per change in planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.